CLINICAL TRIAL: NCT02307643
Title: An Exploratory Study of MT-1303 in Subjects With Systemic Lupus Erythematosus (a Multicenter, Open-label Study)
Brief Title: Exploratory Study of MT-1303 in Systemic Lupus Erythematosus Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tanabe Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MT-1303-J03
Record Dates: First submitted 2014-11-18; First posted 2014-12-04 (Estimated); Last update posted 2017-06-14 (Actual); Status verified 2017-06

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Systemic lupus erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — amiselimod

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Part 1 (Experimental): MT-1303 Low dose+Corticosteroid
  Interventions: Drug: MT-1303 Low dose
- Part 2-A (Experimental): MT-1303 High dose+Corticosteroid
  Interventions: Drug: MT-1303 High dose
- Part 2-B (Experimental): MT-1303 Low dose+Corticosteroid+Immunosuppressant
  Interventions: Drug: MT-1303 Low dose

INTERVENTIONS:
Drug: MT-1303 Low dose
  Arms: Part 1; Part 2-B
Drug: MT-1303 High dose
  Arms: Part 2-A

SUMMARY:
The purpose of this study is to evaluate the safety/tolerability and to explore the efficacy of MT-1303 in subjects with systemic lupus erythematosus

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of SLE based on the American College of Rheumatology (ACR) criteria
* Presence of at least one of the following items: positive anti ds-DNA antibodies, low complement levels, and so on.
* Stable doses of corticosteroids

Exclusion Criteria:

* Severe active lupus nephritis, neuropsychiatric SLE

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2015-02; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Number of Subjects with Adverse Events | up to 36 weeks

SECONDARY OUTCOMES:
Change from Baseline in anti-dsDNA and complement | baseline and 24 weeks
Change from Baseline in Lymphocyte counts | baseline and 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Tsutomu Takeuchi, MD, Study Chair — Keio University Hospital; Yoshiya Tanaka, MD, Study Director — University of Occupational and Environmental Health; Kazuoki Kondo, MD, Study Director — Tanabe Pharma Corporation
Locations (14):
- Japan (14):
  - Inverstigational site, Bunkyō City
  - Inverstigational site, Chiba
  - Inverstigational site, Chūōku
  - Inverstigational site, Fuchu-shi
  - Investigational site, Fukuoka
  - Inverstigational site, Kawagoe-shi
  - Inverstigational site, Maebashi
  - Inverstigational site, Meguro-ku
  - Investigational site, Narashino-shi
  - Investigational site, Sendai
  - Inverstigational site, Shimotsuga-gun
  - Inverstigational site, Shinjuku-ku
  - Inverstigational site, Tsukuba
  - Investigational site, Urayasu-shi

REFERENCES:
- [Derived] Tanaka Y, Kondo K, Ichibori A, Yanai Y, Susuta Y, Inoue S, Takeuchi T. Amiselimod, a sphingosine 1-phosphate receptor-1 modulator, for systemic lupus erythematosus: A multicenter, open-label exploratory study. Lupus. 2020 Dec;29(14):1902-1913. doi: 10.1177/0961203320966385. Epub 2020 Oct 28. PMID 33115374